CLINICAL TRIAL: NCT05297253
Title: Prosthetic and Biological Complications of Implant Retained Fixed Versus Removable Telescopic Overdentures
Brief Title: Prosthetic and Biological Complications of Implant Supported Prostheses
Status: Completed | Type: Observational
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Eman Gamal Helal, Doctor, National Research Centre, Egypt
Other Study IDs: 20199
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Implant Complication
Keywords: dental implant prosthesis; completely edentulous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- telescopic overdenture group: patients receiving implant retained telescopic overdentures
- fixed group: patients receiving fixed implant prostheses
  Interventions: Device: telescopic overdenture

INTERVENTIONS:
Device: telescopic overdenture — fixed implant retained prostheses
  Other Names: fixed implant prosthses
  Groups: fixed group

SUMMARY:
complications of implant retained prostheses

DETAILED DESCRIPTION:
counting and analyzing the prosthetic and biological complications of the fixed and removable implant retained prostheses in the completely edentulous patients

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patients

Exclusion Criteria:

* medically free adequate bone quality and quantity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: completely edentulous patients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
biological complications | one month
  biological complications of implant retained prostheses

SECONDARY OUTCOMES:
prosthetic complications | three months after delivery of the prostheses
  prosthetic complications of implant retained prostheses

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided